CLINICAL TRIAL: NCT03893890
Title: A Phase 2b, Open Label Durability Study of EN3835 Following Treatment of Edematous Fibrosclerotic Panniculopathy
Brief Title: Durability and Safety of EN3835 in the Treatment of EFP (Cellulite) in Women
Status: Completed | Type: Observational
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: EN3835-219
Record Dates: First submitted 2019-02-15; First posted 2019-03-28 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Edematous Fibrosclerotic Panniculopathy
Keywords: Edematous Fibrosclerotic Panniculopathy; EFP; Cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No Treatment: Subjects who participated in and completed studies EN3835-201 and EN3835-202 and had composite improvement of at least 2 levels on both the CR-PCSS and PR-PCSS in the EN3835-201 study, will be eligible for this study. The study will consist of up to two evaluations approximately 3 years after the first dose of study drug was received in the EN3835-201 study.
  Interventions: Biological: Previously Treated with EN3835

INTERVENTIONS:
Biological: Previously Treated with EN3835 — No treatment to be administered - Observational only

SUMMARY:
This is a Phase 2b, rollover, long-term study to evaluate the safety and duration of efficacy of EN3835 in the treatment of women with EFP. Subjects who participated in and completed studies EN3835-201 and EN3835-202 and had composite improvement of at least 2 levels on both the CR-PCSS and PR-PCSS in study EN3835-201 will be eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

* To qualify for the study a subject must:

  1. Be able to provide voluntary written informed consent prior to the initiation of any study-specific procedures per the policy of the governing Institutional Review Board (IRB)/Independent Ethics Committee (IEC).
  2. Have participated in and completed both studies EN3835-201 and EN3835-202 and had composite improvement of at least 2 levels on both the CR-PCSS and PR-PCSS in study EN3835-201.
  3. Be willing and able to comply with all protocol required visits and assessments.

Exclusion Criteria:

* Subjects will be ineligible for participation in this study if the subject:

  1. Has had retreatment with EN3835 in the area initially treated during the EN3835-201 study since the completion of study EN3835-202.
  2. Has had liposuction on the body region treated during the EN3835-201 study since the completion of that study.
  3. Has had any of the following in the area initially treated during the EN3835-201 study since the completion of that study.

     1. Injections (eg, mesotherapy); radiofrequency device treatments; laser treatment; or surgery (including subcision and/or powered subcision).
     2. Any investigational treatment for EFP/cellulite.
     3. Endermologie® or similar treatments.
     4. Massage therapy.
     5. Creams (eg, Celluvera™, TriLastin®).
  4. Any other condition(s) that, in the Investigator's opinion, might indicate the subject is unsuitable for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Up to 8 subjects who completed the EN3835-201 and EN3835-202 studies and who had a composite improvement of at least 2 levels on both the CR-PCSS and PR-PCSS in the EN3835-201 study.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline of response to treatment with EN3835 in subjects with EFP as assessed using the Clinician Reported Photonumeric Cellulite Severity Scale (CR-PCSS) | Change from baseline (pre-dose, Day 1) of response to treatment, approximately 3 years post treatment in EN3835-201 Study
  Change from baseline (pre-dose, Day 1) of EN3835-201 study in CR-PCSS Scale is 5-levels, 0=None to 4=Severe
Change from baseline of response to treatment with EN3835 in subjects with EFP as assessed using the Patient Reported Photonumeric Cellulite Severity Scale (PR-PCSS) | Change from baseline (pre-dose, Day 1) of response to treatment, approximately 3 years post treatment in EN3835-201 Study
  Change from baseline (pre-dose, Day 1) of EN3835-201 study in PR-PCSS Scale is 5-levels, 0=None to 4=Severe
Change from reference time point of response to treatment with EN3835 in subjects with EFP as assessed using the Clinician Reported Photonumeric Cellulite Severity Scale (CR-PCSS) | Change from reference time point (Day 71), approximately 3 years post treatment in EN3835-201 Study
  Change from reference time point (Day 71) of EN3835-201 study in CR-PCSS Scale is 5-levels, 0=None to 4=Severe
Change from reference time point of response to treatment with EN3835 in subjects with EFP as assessed using the Patient Reported Photonumeric Cellulite Severity Scale (PR-PCSS) | Change from reference time point (Day 71), approximately 3 years post treatment in EN3835-201 Study
  Change from reference time point (Day 71) of EN3835-201 study in PR-PCSS Scale is 5-levels, 0=None to 4=Severe

CONTACTS AND LOCATIONS:
Overall Officials: Karen Chajko, Study Director — Endo Pharmaceuticals
Locations (5):
- United States (5):
  - Endo Clinical Trial Site #4, Clearwater, Florida
  - Endo Clinical Trial Site #1, Coral Gables, Florida
  - Endo Clinical Trial Site #5, Washington, Missouri
  - Endo Clinical Trial Site #2, New York, New York
  - Endo Clinical Trial Site #3, Charlottesville, Virginia